CLINICAL TRIAL: NCT02370225
Title: Effects of Aerobic Exercise on Fatigue in Women With Primary Sjögren's Syndrome: Randomized Controlled Trial
Brief Title: Aerobic Exercise in Primary Sjögren's Syndrome
Acronym: AEPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samira Tatiyama Miyamoto (Other)
Collaborators: Federal University of São Paulo (Other); Newcastle University (Other)
Responsible Party: Sponsor-Investigator, Samira Tatiyama Miyamoto, Prof MSc, Federal University of Espirito Santo
Organization: Federal University of Espirito Santo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRPPG 3363/2012
Record Dates: First submitted 2015-02-09; First posted 2015-02-24 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Sjogren's Syndrome
Keywords: sjogren's syndrome; aerobic exercise; fatigue
MeSH Terms: conditions — Sjogren's Syndrome; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic exercise (Experimental): Subjects were submitted to a supervised walking, 3 times a week for 16 weeks.
  Interventions: Other: aerobic exercise
- no exercise (No Intervention): Subjects randomized to control group did not participate of the walking exercise initially, but after completing 16 weeks they were invited to participate of the training group.

INTERVENTIONS:
Other: aerobic exercise — Each training session was preceded by a warm-up period, where patients were instructed to walk freely and slowly for 5 minutes, followed by 20 to 50 minutes of effective walking when they were instructed to maintain their paces to achieve the target heart rate and ending by a cold-up period for 5 minutes (similar to warm-up period).
  The exercise prescription was based on the heart rate at the anaerobic threshold determined at the initial assessment. The increment of intensity exercise was based on time: 30 in the first 2 weeks, adding 5 minutes per week until eighth week, completing 60 minutes, which remains until the end.
  Arms: aerobic exercise

SUMMARY:
The purpose of this sudy is to investigate the effects of a regular aerobic exercise on aerobic capacity, fatigue, depression, quality of life, perception of symptoms and disease activity in women with pSS.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. 45 women with primary Sjögren's syndrome diagnosed according to the American European Consensus Criteria (VITALI et al, 2002) and age ≤ 65 years-old will be included. Patients, in blocks of four, will be allocated to treatment group (TG) or control group (CG) by simple randomization according to drawing lots.

Treatment group (TG): subjects will be submitted to a supervised walking, 3 times a week for 16 weeks, by one physiotherapist and one physical education student who alternated weekly. The heart rate of the patients will be registered with a pulse watch (Polar® A1, Kempele, Finland) at the beginning, in the intermediate time and at the final of effective walking time. The general exertion was rated on the Borg RPE 0-10 (ratings of perceived exertion) scale in the intermediate time and at the final of effective walking time. Each training session will be preceded by a warm-up period, where patients will be instructed to walk freely and slowly for 5 minutes, followed by 20 to 50 minutes of effective walking when they will be instructed to maintain their paces to achieve the target heart rate and ending by a cold-up period for 5 minutes (similar to warm-up period).

The exercise prescription will be based on the heart rate at the anaerobic threshold determined at the initial assessment according previous studies with patients with fibromyalgia (VALIM et al, 2002; VALIM et al, 2003; ASSIS et al, 2006) and Systemic Lupus Erythematosus (CARVALHO et al, 2005), which demonstrated that ventilatory anaerobic threshold oxygen uptake, although used less than VO2max, is also a good physical fitness indicator, and it has the advantage of not being maximum effort dependent. It seems to be more influenced by training than VO2max and represents a safer intensity for exercise, thus decreasing the risk of lesions and constituting an important measure for prescription of exercise. As there is no previous studies using spiroergometric test in pSS and fatigue is very similar to fibromyalgia and lupus patients, we believe pSS performance in treadmill test and training is probably the same. The increment of intensity exercise will be based on time: 30 in the first 2 weeks, adding 5 minutes per week until eighth week, completing 60 minutes, which remains until the end.

Control group (CG): subjects randomized to control group will not participate of the walking exercise initially, but after completing 16 weeks they will be invited to participate of the training group.

Clinical outcomes:

* Fatigue: Functional Assessment of Chronic Illness Therapy Fatigue Subscale (FACIT-Fatigue) (WEBSTER et al, 1999; WEBSTER et al, 2003)
* Depression: Beck Depression Inventory (BDI) (BECK et al, 1961; GORESTEIN and ANDRADE, 1996).
* Perception of pSS's symptoms: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) (SEROR et al, 2011, PAGANOTTI et al, 2012; PAGANOTTI et al, 2013).
* Disease activity: EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) (SEROR et al, 2010; SERRANO et al, 2013).
* Quality of life: Medical Outcomes Study 36 (SF-36) (CICONELLI et al, 1999) and World Health Organization Quality of Life Instrument - Abbreviated version (WHOQOL-bref) (The Whoqol Group, 1998; FLERCK et al, 2000).
* All patients will be submitted to interview to evaluate fatigue, depression and perception of pSS's symptoms prior to intervention (T0), after 8 weeks (T1) and after 16 weeks (T2). Quality of life and disease activity will be evaluated prior to intervention (T0) and after 16 weeks (T2). Patient global assessment of response to therapy (PGART) on a 5-point scale (1 _ much better, 2 _ better, 3 _ slightly better, 4 _ no change, and 5 _ worse).

Physical fitness outcomes:

Aerobic capacity will be evaluated by spiroergometric test. A computerized metabolic system is used to analyze the data obtained breath by breath. The following outcomes of physical fitness are obtained: peak oxygen uptake (peak VO2), peak heart rate and maximum heart rate at the anaerobic threshold. Anaerobic threshold are considered the mean value of 2 blinded investigators' independent readings. Considering that patients with pSS do not achieve a maximum effort, the anaerobic threshold is the main measure of aerobic fitness (VALIM et al, 2002; VALIM et al, 2003; ASSIS et al, 2006).

All the patients will be underwent an increasing load protocol on the treadmill, with a maximum duration of 13 minutes (VALIM et al, 2002; FAIRSHTER et al, 1983). Beginning with a warm-up period of 3 minutes at 3 km/h and increasing 1 km/h each minute until 7 km/h, at this moment 2,5% inclination is added until 15% in the 13º minute.

All patients will be evaluated prior to intervention (T0) and after 16 weeks (T2).

Statistics:

An intent-to-treat analysis will be performed, using the last-observation-carried-forward method. A level of significance of P<0.05 (2-tailed tests) will be accepted for the trial. The Kolmogorov-Smirnov test will be used to determine whether data will be normally or non-normally distributed. For normally distributed data, the dependent variables will be analyzed using a 2 per 3 repeated-measures analysis of variance (ANOVA). The independent variables in all analyses is group (TG versus CG; between subjects factors) and time (baseline, 8 weeks, and 16 weeks; within subjects factors). Independent sample t-tests will be used in the between-groups comparison of the change scores at midline and treatment completion, when interaction time x group was significant. A 95% confidence interval (95% CI) will be used. Friedman's test will be used for non-normally distributed variables, as an equivalent of ANOVA. Wilcoxon's signed rank test will be used to analyze the difference between times separated by group when the change score was non-normally distributed. Fisher's exact test and chisquare test will be used to determine differences in rates of improvement between the 2 groups. Pearson's and Spearman's correlation coefficients will be used. Multiple linear regression and chi-square tests will be used to analyze the association between the amount of physical fitness improvement and outcome measures. The agreement between heart rate and ratings of perceived exertion during the training will be analyzed by Intraclass Correlation Coefficient.

ELIGIBILITY:
Inclusion Criteria:

* female gender and age ≤ 65 years-old
* pSS diagnosed according to the American European Consensus Criteria (VITALI et al, 2002)
* corporal mass index < 40.

Exclusion Criteria:

* use of beta-blocker therapy;
* severe manifestations on pulmonary, renal, neurologic or musculoskeletal system (from the disease or not);
* limiting or hindering their ability to walking performance
* those who had performed regular physical activity in the 6 weeks before trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fatigue at 16 weeks | baseline and 16 weeks
  questionnaires: Functional Assessment of Chronic Illness Therapy Fatigue Subscale (FACIT-Fatigue) (WEBSTER et al, 1999; WEBSTER et al, 2003)

SECONDARY OUTCOMES:
Change from baseline in aerobic capacity at 16 weeks | baseline and 16 weeks
  Aerobic capacity has been evaluated by spiroergometric test. A computerized metabolic system is used to analyze the data obtained breath by breath. The following outcomes of physical fitness are obtained: peak oxygen uptake (peak VO2), peak heart rate and maximum heart rate at the anaerobic threshold. Anaerobic threshold are considered the mean value of 2 blinded investigators' independent readings. Considering that patients with pSS do not achieve a maximum effort, the anaerobic threshold is the main measure of aerobic fitness (VALIM et al, 2002; VALIM et al, 2003; ASSIS et al, 2006).
  All the patients have been underwent an increasing load protocol on the treadmill, with a maximum duration of 13 minutes (VALIM et al, 2002; FAIRSHTER et al, 1983). Beginning with a warm-up period of 3 minutes at 3 km/h and increasing 1 km/h each minute until 7 km/h, at this moment 2,5% inclination is added until 15% in the 13º minute.
Change from baseline in depression at 8 weeks | baseline and 8 weeks
  questionnaire: Beck Depression Inventory (BDI) (BECK et al, 1961; GORESTEIN and ANDRADE, 1996).
Change from baseline in depression at 16 weeks | baseline and 16 weeks
  questionnaire: Beck Depression Inventory (BDI) (BECK et al, 1961; GORESTEIN and ANDRADE, 1996).
Change from baseline in disease activity at 16 weeks | baseline and 16 weeks
  questionnaire: EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) (SEROR et al, 2010; SERRANO et al, 2013).
Change from baseline in quality of life at 16 weeks | baseline and 16 weeks
  questionnaires: Medical Outcomes Study 36 (SF-36) (CICONELLI et al, 1999) and World Health Organization Quality of Life Instrument - Abbreviated version (WHOQOL-bref) (The Whoqol Group, 1998; FLERCK et al, 2000).
Change from baseline in symptoms at 8 weeks | baseline and 8 weeks
  questionnaire: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) (SEROR et al, 2011, PAGANOTTI et al, 2012; PAGANOTTI et al, 2013).
Change from baseline in symptoms at 16 weeks | baseline and 16 weeks
  questionnaire: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) (SEROR et al, 2011, PAGANOTTI et al, 2012; PAGANOTTI et al, 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, PhD, Study Chair — Universidade Federal de São Paulo
Locations (1):
- Samira Tatiyama Miyamoto, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miyamoto ST, Valim V, Carletti L, Ng WF, Perez AJ, Lendrem DW, Trennel M, Giovelli RA, Dias LH, Serrano EV, Subtil AM, Abreu VC, Natour J. Supervised walking improves cardiorespiratory fitness, exercise tolerance, and fatigue in women with primary Sjogren's syndrome: a randomized-controlled trial. Rheumatol Int. 2019 Feb;39(2):227-238. doi: 10.1007/s00296-018-4213-z. Epub 2019 Jan 2. PMID 30604204